CLINICAL TRIAL: NCT04300803
Title: An Expanded Access Protocol to Provide Intermediate Access to Tafasitamab (MOR208) for the Combination Treatment With Lenalidomide to Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL)
Brief Title: Expanded Access Program for Tafasitamab (MOR00208) in R/R DLBCL
Status: Approved for marketing | Type: Expanded Access
Sponsor: MorphoSys AG (Industry)
Collaborators: Clinigen Healthcare Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: MOR208N001
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-05

CONDITIONS: DLBCL
Keywords: Tafasitamab; MOR00208; MOR208; monoclonal anti-CD19 antibody; Diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Tafasitamab, 12 mg/kg. 4 week cycles: weekly (Cycle 1-3) to bi-weekly (Cycle 4 onwards), loading dose Cycle 1, day 4. Cycle 4 onwards day 1, day 15 until disease progression — Expanded Access Program, Non-Interventional Study

SUMMARY:
Expanded Access Program (EAP) to provide Tafasitamab (MOR208) to eligible patients with relapsed or refractory Diffuse Large B Cell Lymphoma. Access to MorphoSys´ EAP can be requested by contacting the respective CRO Clinigen (tafasitamab@clinigengroup.com).

DETAILED DESCRIPTION:
This program is intended to provide access to patients with relapsed and/or refractory DLBCL who had at least one prior anti-CD20 containing regimen. Patients with primary refractory disease and double/triple hit status are also eligible. Patients considering this access program should have no other therapeutic option, and are not eligible for other clinical trials. The expanded access program (MOR208N001) is currently available in the United States only.

ELIGIBILITY:
Major Inclusion Criteria :

1. Age ≥ 18 years
2. Patient able to provide written informed consent
3. Histologically-confirmed diagnosis of DLBCL, including transformation from an earlier diagnosis of indolent lymphoma.
4. Patients must have relapsed and/or refractory DLBCL, including primary refractory disease and double/triple hit status, after at least 1 prior anti-CD20 containing regimen.
5. Patients with a serious, life-threatening illness in which conventional therapies have failed, are unsuitable and/or are unavailable and participation in ongoing relevant clinical trials is not feasible.

Major Exclusion Criteria:

1. Patients who have other histological type of lymphoma, e.g. indolent Non-Hodgkin lymphoma (NHL), Primary mediastinal B-cell lymphoma (PMBL) or Burkitt Lymphoma
2. Patients who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period with lenalidomide
3. Patients with:

   1. Known active bacterial and viral and fungal infections
   2. Serology of chronic active viral Hepatitis B and/or C-Hepatitis
   3. Known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV)
4. Patients who are unable to participate in the lenalidomide REMS program

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult